CLINICAL TRIAL: NCT06458166
Title: Associations Between Low Frequency Fatigue, Jump Height and Perceptual Measures of Muscle Soreness, Fatigue and Recovery in Youth Elite Soccer Players
Brief Title: Associations Between Low Frequency Fatigue, Jump Height and Perceptual Measures of Muscle Soreness, Fatigue and Recovery
Status: Recruiting | Type: Observational
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Other Study IDs: ST_S_
Record Dates: First submitted 2024-06-01; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Fatigue; Physical Exercise
Keywords: sports; soccer; low frequency fatigue
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of low frequency fatigue using low frequency eletrical stimulation — Pre-programmed muscle electrical stimuli will be applied via Myocene® software using 3 electrodes: 1 cathode (5 x 10 cm) placed transversely over the proximal quadriceps femoris, and 2 anodes (5 x 5 cm) over the distal vastus medialis and vastus lateralis. Sixteen sets of stimuli will be administered with 5 seconds between sets. Each set consists of a single pulse, a train of 5 stimuli at 20 Hz, and a train of 18 stimuli at 120 Hz, with 1-second intervals between. The stimulation intensity starts at 25 mA and increases by 1 mA per set, reaching 40 mA in the final set. The Myocene® software calculates the ratio of low- to high-frequency evoked forces within each set. The outcome (Powerdex) is the median value of these 16 ratios for each leg. This evaluation will be conducted on both legs, taking 2 minutes per leg.

SUMMARY:
Over the recent years, the increased competitive demands in elite competitive athletes has sparked a heightened interest in monitoring fatigue. Given the nature of the soccer game, athletes may experience low-frequency fatigue. Until recently, this assessment was restricted to in-lab. However, the emergence of new instruments aiming to allow low-frequency assessment to be carried out on a daily basis, in the context of professional teams. This study aimed to analyze the recovery of low-frequency fatigue, jump height and perceptual responses following competition and investigate possible associations between the objective and subjective parameters.

ELIGIBILITY:
Inclusion Criteria:

* Elite level youth soccer players, competing in the highest portuguese division

Exclusion Criteria:

* Older adults
* none elite soccer player
* Play less than 70 minutes of match

Ages: 16 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Players at the highest division of the portuguese national championships in their respective age group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-21 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences in Low frequency fatigue measured using Myocene (eletrical stimulus and force measurement) | 2 hours before the match; 30 minutes following the match, 24 hours following the match; 48 hours following the match
  Assessment using myocene. Muscles are stimulated with low-frequency electrical pulses. The response of the muscle (force or torque) output, is recorded. A decrease in force output compared to baseline levels indicates fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided